CLINICAL TRIAL: NCT02221050
Title: Influence of Chronic Renal Failure and Hemodialysis on Liking and Wanting for Foods
Brief Title: Hemodialysis and Wanting for Protein-rich Foods
Status: Completed | Type: Observational
Sponsor: University of Burgundy (Other)
Responsible Party: Principal Investigator, Laurent BRONDEL, University professor, University of Burgundy
Other Study IDs: 2013/28
Record Dates: First submitted 2014-08-13; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
A study conducted in the laboratory revealed the existence of a "window" during which patients with renal failure appreciate the protein-rich foods. This period, located immediately after the dialysis, is likely related to the purification of plasma products resulting from protein catabolism. It therefore appears necessary to understand the mechanisms that may explain these changes by measurements of ghrelin (orexigenic hormone), leptin (anorectic hormone) and plasma amino acids.

DETAILED DESCRIPTION:
In 24 patients with renal failure treated by hemodialysis, it is evaluated (at 8:00 am and at 11:00 am), a day without hemodialysis and another day after the hemodialysis:

* Hunger sensation,
* Olfactory liking assessed separately for 6 foods (2 carbohydrate-, 2 fat- and 2 protein-rich foods) and 2 non-alimentary products,
* Food wanting evaluated by the sequential presentation of 18 images of food (6 fat-, 6 carbohydrate- and 6 protein-rich foods),
* Two blood samples for the assays of leptin, ghrelin, creatinine, albumin and pre-albumin as well as plasma amino acids.

  24 healthy subjects are also evaluated in order to compare the results from patients to those of control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients and healthy subjects were included if they were aged between 18 and 80 years

Exclusion Criteria:

* diabetes, advanced undernutrition (BMI < 17.5 kg m-2, prealbumin < 250 mg.L-1), congestive heart failure, acute or chronic infection, ongoing antibiotic treatment, active cancer, liver cirrhosis, smoking (more than 5 cigarettes/day), alcohol consumption (more than 3 units/day), aversion to the foods eaten or smelt during the study, impaired comprehension of the cognitive tasks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hemodialysis centers of Clinique Drevon, Dijon, France la Breuchillière, Saint Apollinaire, France University Hospital, Dijon, France Macon Hospital, Macon, France
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Amount of wanting for protein-rich foods | 20 min (from 8:00 to 8:20 am) and 20 min (from 11:00 to 11:20 am)
  The wanting is determined after the successive presentation (for ten seconds) of 18 pictures of food. For each food the question is "at the present time, do you want to eat this food? ". For each photo, subjects place a vertical line on a 10 cm horizontal line bounded at its ends by "no desire" and "extremely envy" (visual analog scale).The wanting for proteins is the mean score for the desire to eat protein-rich foods.

SECONDARY OUTCOMES:
Concentrations of the plasma amino-acids | 8:30 am and 11:30 am
  Variation in concentrations of amino-acids during the morning a day with hemodialysis and a day without hemodialysis, and comparison with plasma AAs from healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Luc PENICAUD, PHD, Study Director — Centre des Sciences du Goût, Centre National de la recherche Scientifique
Locations (1):
- Centre des Sciences du Goût, Dijon, Burgundy, France

REFERENCES:
- [Derived] Mouillot T, Filancia A, Boirie Y, Brindisi MC, Hafnaoui N, Van Wymelbeke V, Teillet E, Meintani I, Jacquin-Piques A, Leloup C, Penicaud L, Mousson C, Brondel L. Hemodialysis Affects Wanting and Spontaneous Intake of Protein-Rich Foods in Chronic Kidney Disease Patients. J Ren Nutr. 2021 Mar;31(2):164-176. doi: 10.1053/j.jrn.2020.05.006. Epub 2020 Jul 25. PMID 32723525